CLINICAL TRIAL: NCT00811447
Title: Open Label, Randomized Multicenter Study Docetaxel + 5-fluorouracil + Cisplatin Compared to Cisplatin + 5-fluorouracil in Patients With Metastatic or Locally Recurrent Gastric Cancer Previously Untreated With Chemotherapy for Advanced Disease
Brief Title: Taxotere New Indication - Gastric Cancer Treatment Registration Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_02195
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2012-08-31 (Estimated); Status verified 2012-08

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Fluorouracil; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Administration of docetaxel 60 mg/m² on Day 1, Cisplatin 60 mg/m² after the end of the docetaxel infusion and 5-fluorouracil (5-FU) 600 mg/m²/day from Day 1 after the end of the cisplatin infusion to Day 5.
  Interventions: Drug: 5-fluorouracil; Drug: Cisplatin; Drug: Docetaxel
- 2 (Active Comparator): Cisplatin 75 mg/m² on Day 1, 5-FU 600 mg/m²/day from Day 1 after the end of the cisplatin infusion to Day 5.
  Interventions: Drug: 5-fluorouracil; Drug: Cisplatin

INTERVENTIONS:
Drug: 5-fluorouracil — 600 mg/m²/day intravenous
Drug: Cisplatin — 60 mg/m² or 75 mg/m² intravenous
Drug: Docetaxel — 60 mg/m² intravenous
  Arms: 1

SUMMARY:
Primary objective:

To detect a statistically significant increase in time to progression (TTP) of disease for the test group (Taxotere® [Docetaxel] combined with cisplatin and 5-fluorouracil [TCF]) relative to the control group (Cisplatin combined with 5-fluorouracil[CF])

Secondary objectives:

* To detect a statistically significant increase in overall survival (OS) for the test group relative to the control group.
* To compare response rate (RR), time to treatment failure (TTF), duration of responses, safety profiles, quality of life (QOL), and disease-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma including adenocarcinoma of the esophagogastric junction, histologically proven.
* Measurable and/or evaluable metastatic disease; if a single metastatic lesion is the only manifestation of the disease, cytology or histology is mandatory. Locally recurrent disease is accepted provided that there is at least one measurable lesion.
* Performance status Karnofsky index >70%
* Life expectancy of more than 3 months
* Adequate haematological parameters (Hb≥9g/dl, ANC≥2.0× 109/L, platelets ≥ 100× 109/L)
* Creatinine ≤ 1.25 UNL, serum magnesium should be within the normal value
* Total bilirubin ≤ 1 UNL, AST and ALT ≤ 2.5 UNL, alkaline phosphatase ≤ 5 UNL
* No prior palliative chemotherapy, previous adjuvant chemotherapy is allowed if more than 12 months has elapsed between the end of adjuvant therapy and first relapse.
* At least 6 weeks from prior radiotherapy and 3 weeks from surgery
* Complete initial work-up within two weeks prior to first infusion for clinical evaluation and biological work-up. Abdominal CT scan and chest X-rays are mandatory.

Exclusion Criteria:

* Pregnant or lactating women
* Patients with reproductive potential not implementing adequate contraceptive measures
* Other tumor type than adenocarcinoma
* Any prior palliative chemotherapy. Prior adjuvant chemotherapy with a first relapse within 12 months from the end of adjuvant
* Prior treatment with taxanes. Prior CDDP as adjuvant chemotherapy with cumulative dose > 300mg/m²
* Previous or current malignancies other than gastric carcinoma, with the exception of adequately treated in situ carcinoma of the cervix uteri or non melanoma skin cancer
* Patients with known brain or leptomeningeal metastases
* Symptomatic peripheral neuropathy ≥ grade 2 by NCIC-CTG criteria
* Other serious illness or medical conditions:

  * unstable cardiac disease despite treatment, myocardial infarction within 6 months prior to study entry
  * history of significant neurologic or psychiatric disorders including dementia or seizures
  * active uncontrolled infection
  * active disseminated intravascular coagulation
  * other serious underlying medical conditions which could impair the ability of the patient to participate in the study
* Concurrent treatment with corticosteroids except as use for the prophylactic medication regimen, treatment of acute hypersensitivity reactions or unless chronic treatment at low doses
* Definite contraindications for the use of corticosteroids
* Hypercalcemia not controlled by bisphosphonates and more than 12mg/100ml
* Liver impairment with AST or ALT more than 1.5UNL associated with alkaline phosphatase more than 2.5UNL
* Concurrent or within 4 week period administration of any other experimental drugs
* Concurrent treatment with any other anti-cancer therapy

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2008-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Time to progression | Throughout the study period

SECONDARY OUTCOMES:
Safety profile | Throughout the study period
Overall survival | From beginning to end of study
Tumor response | every 8 weeks
Clinical toxicities/symptomatology | Throughout the study period
Laboratory toxicities/symptomatology | Throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Martin Thoenes, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China